CLINICAL TRIAL: NCT00483964
Title: A Randomized, Controlled ,Clinical Trial of a Herbal Combination of Aqueous Extracts of Bacopa Monnieri and Nardostachys Jatamansi in the Treatment of Schizophrenia, Compared to Standard Anti-Psychotic Drugs
Brief Title: A Safety and Efficacy Study of Bacopa Monnieri and Nardostachys Jatamansi to Treat Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Q.Mundewadi Ayurvedic Research & Charitable Trust (Other)
Collaborators: Stanley Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMRI #04T-512
Record Dates: First submitted 2007-06-06; First posted 2007-06-08 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Herbal extracts; Randomized; Controlled; Clinical Trial
MeSH Terms: conditions — Schizophrenia | interventions — Valeriana extract; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): The group getting the study drugs, Bacopa monnieri and Nardostachys jatamansi
  Interventions: Drug: Bacopa monnieri; Drug: Nardostachys jatamansi
- B (Active Comparator): The group getting Olanzapine
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Bacopa monnieri
  Arms: A
Drug: Nardostachys jatamansi
  Arms: A
Drug: Olanzapine
  Arms: B

SUMMARY:
The purpose of this study is to determine whether a herbal combination of water based extracts of Bacopa monnieri(BM) and Nardostachys jatamansi(NJ) is effective in the treatment of Schizophrenia.

The working hypothesis for this study is that a herbal combination of BM and NJ will be as effective as modern anti-psychotic drugs, in the treatment of Schizophrenia, and will be safe for long term use.

DETAILED DESCRIPTION:
At present, there is no clearly effective treatment of Schizophrenia, which is present in 1% of the population. While acute psychotic episodes are well-controlled with modern medicines, long-term prognosis in terms of quality of life and productivity remain poor. In India, more than 50% of beds in mental hospitals is taken up by Schizophrenic patients, without much of cost-benefit outcome.In clinical practice, Ayurvedic treatment has proved to be effective and well-accepted in patients of Schizophrenia, is safe on long-term use, and may bring about the desired long-term positive changes in patient-health outcome.

In this proposed project, 200 patients of Schizophrenia will be recruited from the local and regional psychiatric institutions. The patients will be in the age group from 18-60 and of either sex. Patients suffering from any organic disorder will not be included in the study. Patients having any concomitant drug addiction will also not be included. Each patient and a close relative (as guardian) will be required to sign a consent form, for the clinical trial, in the regional language. Full, written information about the proposed clinical trial will be given to the patient and relatives. All information will be available in English and two regional languages, viz. Hindi and Marathi. Full detailed history and clinical examination of all patients will be done. Each patient will be interviewed with the Structured Clinical Interview for Axis I DSM-IV Disorders (SCID).Diagnosis of Schizophrenia will be done using the DSM-IV-TR diagnostic criteria for Schizophrenia (from American Psychiatric Association:- Diagnostic and Statistical Manual of Mental Disorders - 2000). This will also include classification of longitudinal course in patients having more than 1 year's duration of onset of active-phase symptoms. The clinical profile of each patient will be evaluated using the Positive and Negative Symptom scale for Schizophrenia. This is a structured clinical interview (SCI-PANSS) having 30 items which rate along a seven point continuum (1 = absent; 7 = extreme severe). The assessment provides separate scores in nine clinical domains including a positive syndrome, a negative syndrome, depression, a composite index, and general psychopathology. The SCI-PANSS will be used for each patient initially for baseline evaluation before commencing treatment and later, once in 3 months, to provide assessment of treatment response. The patients will be divided at random into 2 groups of 100 each, one a study group and the other a control group. A brief wash-out period of 2 weeks will be given to patients already taking some medication. The study group will be given Ayurvedic medicine in the dose of 2 tablets b.i.d. of BM, and 1tablet b.i.d. of NJ; with each 350 mg. tablet containing 200mg of aqueous extract . This dosage is in accordance with prevalent use of the above two herbs, in adults. The control group will be given a standard anti-psychotic drug Olanzapine, 10 mg. o.d.

Patients will be dispensed Ayurvedic medicine or anti-psychotic for 4 weeks and then reassessed at every visit. Basic clinical examination and clinical changes will be noted. Baseline SGPT/B. Urea/ S. Creatinine will be done for all patients and repeated every 6 months, to assess any possible drug toxicity. The progress of the patients will be carefully monitored for a total period of 78 weeks each, with a watch for any possible signs of drugs toxicity, treatment failure or aggravation of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Any sex
* Age 18 - 60 years
* History suggestive of Schizophrenia using the DSM-IV-TR diagnostic criteria.
* Presence of a caretaker/legal guardian who would take the responsibility of giving regular medication and bringing the patient for regular follow-ups.

Exclusion Criteria:

* Age< 18 or > 60 years
* Known history of drug addiction
* Known medical history which may cause similar symptoms e.g. Schizoaffective /Mood Disorders, Pervasive Developmental Disorder
* History of severe or repeated episodes of violence.
* History of any other concurrent illness which could interfere in the treatment and assessment of the subject.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2005-09; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The change in the total PANSS score from baseline till the end of the study. | 78 weeks

SECONDARY OUTCOMES:
The change in physical , clinical , and hematological parameters from baseline till the end of 78 weeks of treatment | 78 weeks

CONTACTS AND LOCATIONS:
Overall Officials: AbdulMubeen A Mundewadi, B.A.M.S., Principal Investigator — Q.Mundewadi Ayurvedic Research & Charitable Trust
Locations (1):
- Q.Mundewadi Ayurvedic Research & Charitable Trust, Mumbra,Thane, Maharashtra, India